CLINICAL TRIAL: NCT06860620
Title: Efficacy of Zinc Supplementation in Maintaining Sustained Remission in Children With Steroid-sensitive Nephrotic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEDNEFMULTAN
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Steroid-Sensitive Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc supplementation plus standard treatment group (Experimental): Children were given 5 mg of elemental zinc sulfate as a single daily dose for children less than 4 years of age and 10 mg for children more than 4 years of age for a total duration of 6 months, along with standard therapy.
  Interventions: Drug: Zinc supplementation plus standard treatment
- Standard treatment (No Intervention): Children received prednisolone at a dose of 60 mg/m2 per day for 4-8 weeks or less if they reached absence of proteinuria for 3 consecutive days, followed by 40 mg/m2 on alternate days for 2 weeks, followed by gradual tapering over 1-2 months to the minimum dose of 0.5 to 1 mg/kg/day for a total duration of 6 months.

INTERVENTIONS:
Drug: Zinc supplementation plus standard treatment — children were given 5 mg of elemental zinc sulfate as a single daily dose for children less than 4 years of age and 10 mg for children more than 4 years of age for a total duration of 6 months, along with standard therapy.
  Arms: Zinc supplementation plus standard treatment group

SUMMARY:
This study aims to fill the gaps by determining the efficacy of zinc supplementation in maintaining sustained remission in children with steroid sensitive nephrotic syndrome (SSNS).

DETAILED DESCRIPTION:
There is a need to ascertain the efficacy of zinc supplementation in maintaining sustained remission in children with SSNS, thereby lowering the number of relapses and disease morbidity. The findings of this study could pave the way for reasonable evidence about the role of zinc supplementation is sustained remission in children with SSNS.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Aged 2-12 years
* With steroid-sensitive nephrotic syndrome, with frequent relapses

Exclusion Criteria:

* Children with steroid-resistant nephrotic syndrome
* With a history of chronic systemic illness (cardiac, metabolic, malignancy, pulmonary, neurologic, or rheumatologic)
* With a history of kidney disease like polycystic kidney disease

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Sustained remission | 6 months
  Efficacy yes if sustained remission was seen after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Saleem, FCPS, Principal Investigator — Nishter Hospital Multan, Pakistan; Afsheen Asghar, FCPS, Principal Investigator — Nishter Hospital Multan, Pakistan; Sheeba Yousuf, FCPS, Principal Investigator — Nishter Hospital Multan, Pakistan
Locations (1):
- Nishtar Hospital, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.